CLINICAL TRIAL: NCT06133777
Title: Description of Respiratory Variability and Postoperative Complications During Thoracic Lung Resection - Exploratory Study.
Brief Title: Respiratory Variability and Postoperative Complications During Thoracic Lung Resection.
Acronym: RESPIVARIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A00931-44
Record Dates: First submitted 2023-10-23; First posted 2023-11-15 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Lung Injury
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory Variability Monitoring (Experimental): Respiratory variability will be measured using a belt equipped with an external sensor allowing automatic and continuous analysis of thoracic movement by frequency analysis
  Interventions: Other: Respiratory variability monitoring

INTERVENTIONS:
Other: Respiratory variability monitoring — Respiratory variability will be measured using a belt equipped with an external sensor allowing automatic and continuous analysis of thoracic movement by frequency analysis

SUMMARY:
Postoperative respiratory complications (PRC) represent a major public health issue. Majority of PRCs occur once the patient leaves the post-interventional monitoring room.

Identifying patients at risk for PRC is therefore an important step for improving their post-operative care. In this context, any clinical marker making it possible to detect early alteration of the respiratory state in the postoperative phase deserves to be evaluated.

This study is based on the hypothesis that measuring indices of respiratory variability which is synonymous with "good respiratory health" can be part of these markers.

The measurement of respiratory variability will be done in patients with thoracic lung resection surgery before anesthetic induction and in the postoperative phase after extubation. It will be measured using a belt equipped with an external sensor allowing automatic and continuous analysis of thoracic movement by frequency analysis

DETAILED DESCRIPTION:
Postoperative respiratory complications (PRC) represent a major public health issue. By PRC, we mean acute respiratory distress, bronchospasm, pleural effusion, respiratory infection, atelectasis, aspiration pneumonia and pneumothorax.

Postoperative respiratory dysfunction reaches its peak in the 48 hours following surgery. Majority of PRCs therefore occur once the patient leaves the post-interventional monitoring room.

Identifying patients at risk for PRC is an important step for improving their post-operative care. For this, there are predictive scores, notably the ARISCAT score, pre-operatively. However, there are few measurement methods to detect early alteration of the respiratory state in the postoperative phase. Therefore, the physician in charge of the patient is alerted late if the patient deteriorates on the respiratory plan.

In this context, any clinical marker making it possible to detect early alteration of the respiratory state in the postoperative phase deserves to be evaluated. Therefore, this study is based on the hypothesis that measuring indices of respiratory variability can be part of these markers. Consequently, this research which aims to describe these indices of respiratory variability is of major interest.

Respiratory variability is synonymous with "good respiratory health". By the opposite, the reduction of this same variability is pathological and indicates an increase in the level of load imposed on the respiratory system.

The measurement of respiratory variability will be done in patients with thoracic lung resection surgery before anesthetic induction and in the postoperative phase after extubation. It will be measured using a belt equipped with an external sensor allowing automatic and continuous analysis of thoracic movement by frequency analysis

ELIGIBILITY:
Inclusion Criteria:

* Patient, man or woman, who signed informed consent
* Patient older than 18 years old
* Patient admitted for planned thoracic resection surgery (lobectomy, bi-lobectomy, pneumonectomy) whatever the etiology is

Exclusion Criteria:

- None (medical aspects)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Coefficient of variation | Day 1
  Each respiratory cycle is defined by an inspiratory time followed by an expiratory time. Ordinary, it is observed a variability compared to the previous cycle in terms of amplitude and temporality. Coefficient of variation is one of the parameters able to measure this respiratory variability.

CONTACTS AND LOCATIONS:
Overall Officials: Kais BEN HASSEN, MD, Principal Investigator — Hôpital privé de Clairval

IPD SHARING:
Plan to Share IPD: No